CLINICAL TRIAL: NCT03140839
Title: Understanding the Psychological Effects and Mechanisms of Imagery Rescripting for Social Anxiety Disorder: A Controlled Experimental Study
Brief Title: Treating Negative Mental Images and Memories in Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Hebrew University of Jerusalem (Other); University of Toronto (Other); Baycrest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORE # 22071
Record Dates: First submitted 2017-04-21; First posted 2017-05-04 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-10

CONDITIONS: Social Anxiety
MeSH Terms: interventions — Implosive Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of three conditions, either Imaginal Rescripting, Imaginal Exposure, or Supportive Counselling
Who Masked: Participant
Masking Description: Participants will be blind to the condition they receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Imaginal Rescripting (Experimental): Imaginal Rescripting (IR) targets imagery-based mental representations embedded within patients negative autobiographical memories related to social anxiety. In IR, patients progress through 3 distinct phases: (1) They "relive" a past negative event in their imagination, (2) are guided to actively change the original memory in their imagination to create more satisfying outcomes, and (3) relive the memory again while incorporating the new information. The IR intervention will be administered in one 90 minute session.
  Interventions: Behavioral: Imaginal Rescripting
- Imaginal Exposure (Active Comparator): Imaginal Exposure (IE) involves repeatedly "reliving" a negative autobiographical memory related to social anxiety from a first-person perspective and actively considering alternative meanings of the memory, but differs from IR in that the original memory itself is never explicitly modified in any way. The IE intervention will be administered in one 90 minute session.
  Interventions: Behavioral: Imaginal Exposure
- Supportive Counselling (Placebo Comparator): Supportive counselling (SC) provides patients with empathic support regarding a negative autobiographical memory related to social anxiety. The SC condition controls for non-specific clinical factors such as therapeutic attention and alliance. SC will be administered in one 60-90 minute session.
  Interventions: Other: Supportive Counselling

INTERVENTIONS:
Behavioral: Imaginal Rescripting — A stand-alone single session intervention for social anxiety disorder
  Other Names: Imagery Rescripting
  Arms: Imaginal Rescripting
Behavioral: Imaginal Exposure — A stand-alone single session intervention for social anxiety disorder
  Arms: Imaginal Exposure
Other: Supportive Counselling — Non-specific talk therapy focused on non-directive and empathic listening and on supporting patients' existing coping skills and strategies.
  Arms: Supportive Counselling

SUMMARY:
The proposed research will study the effects of Imaginal Rescripting (IR) for social anxiety disorder (SAD). IR guides patients to change their memories of past socially painful events. Initial studies have found that a single session of IR significantly reduces SAD symptoms, however it is not yet clear how or why IR works and whether its effects are long lasting. To answer these questions, the investigators will randomly assign adults with SAD to receive either IR, or two other types of brief psychological interventions: Imaginal Exposure and Supportive Counselling. Changes in participants' memories, social anxiety symptoms, quality of life, negative beliefs, and social behaviour over the course of a 6-month period will be assessed. This study will provide valuable insight into the short- and long-term effects of IR and clarify the mechanisms through which IR works. Ultimately, this knowledge will enable the development of more effective treatments and prevention programs for SAD.

DETAILED DESCRIPTION:
Purpose:

Building upon extensive prior research by the investigators' expert team, the proposed study will examine the effects of Imaginal Rescripting (IR) as a stand-alone single session intervention for social anxiety disorder (SAD). IR is a short but effective cognitive behavioural intervention, which guides patients to change their memories of past socially painful events. The purpose of the study is to examine the effects of IR in relation to two comparison conditions and by doing so also provide much-needed experimental evidence in clinical participants to distinguish between competing theories of treatment mechanisms. Does IR work by altering the content of the memory or simply by changing its meaning or impact, or both? If modifying memory content is important, does IR improve access to more positive memory details that compete with the original negative ones for activation in subsequent contexts or eradicate elements of the original traumatic memory, perhaps via the disruption of memory reconsolidation? The study will take advantage of the recent development and validation of the Waterloo Images and Memories Interview, which enables researchers to measure the accessibility, subjective appraisals, and narrative content of autobiographical memories (and associated mental images) that participants report experiencing. One particularly important outcome generated by the WIMI for the present study involves having trained coders count the number of "episodic" vs. "non-episodic" negative and positive autobiographical memory details present in participants' reported narratives over time.

Research Questions:

The effects of IR will be investigated in comparison to Imaginal Exposure (IE) and Supportive Counselling (SC). IR targets imagery-based mental representations embedded within patients autobiographical memories. In IR, patients progress through 3 distinct phases: (1) Participants "relive" a past negative event in their imagination, (2) are guided to actively change the original memory in their imagination to create more satisfying outcomes, and (3) relive the memory again while incorporating the new information. IE involves repeatedly "reliving" the memory from a first-person perspective and actively considering alternative meanings of the memory, but differs from IR in that the original memory itself is never explicitly modified in any way. SC provides patients with empathic support and controls for non-specific clinical factors such as therapeutic attention and alliance. The research will examine whether IR outperforms these conditions and leads to sustained changes in SAD symptoms, quality of life, and social behaviour. The use of IE as a control condition will help to determine whether the therapeutic effects of IR depend on altering the content of the targeted autobiographical memory rather than just its meaning.

Justification:

Only 3 preliminary studies, including one from the investigators' lab, have examined the effects of IR as a stand-alone intervention for SAD. These studies found that a single 90-min session of IR produced large improvements in SAD symptoms at post-treatment, but both relied exclusively on self-report measures. Moreover, neither study incorporated an active imagery-based control condition against which the specific mechanisms of IR could be experimentally isolated and understood. Understanding the mechanisms of IR will help to facilitate the development of effective treatment and relapse prevention strategies for SAD as well as the future dissemination of efficient but potent CBT interventions to patients diagnosed with SAD.

Objectives:

Capitalizing on innovative methodological advancements in the investigators' lab that enable the precise measurement of patients' memory narratives and appraisals over time, the objective is to elucidate how fear memories are represented in the socially anxious mind, how they change during IR, and how impactful and enduring these effects may be.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of social anxiety disorder (as per DSM-5)
* Endorsement of relevant images/memories associated with social situations.
* Participants currently undergoing stable drug treatment or psychological treatment for anxiety or mood difficulties may be included in the study if the treatment would not interfere with the study interventions.

Exclusion Criteria:

* Active suicidality, psychosis, or an actively-interfering alcohol/substance use disorder.
* Participant does not endorse mental images/memories

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Change in self-reported social anxiety symptoms | Pre-treatment, 1 week, 2 weeks, and 3 months after treatment
  Social Phobia Inventory
Change in clinician-rated social anxiety symptoms | Pre-treatment, 1 week, 2 weeks, and 3 months after treatment
  Liebowitz Social Anxiety Scale-Clinician Rated Version
Change in memory narratives and appraisals | Pre-treatment, 1 week, 2 weeks, and 3 months after treatment
  Waterloo Images and Memories Interview

SECONDARY OUTCOMES:
Change in behavioral indices of social anxiety | Pre-treatment, 1 week, 2 weeks, and 3 months after treatment
  Behavioural Assessment Task
Change in quality of life | Pre-treatment, 1 week, 2 weeks, and 3 months after treatment
  Outcome rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo Department of Psychology and Centre for Mental Health Research, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reimer SG, Moscovitch DA. The impact of imagery rescripting on memory appraisals and core beliefs in social anxiety disorder. Behav Res Ther. 2015 Dec;75:48-59. doi: 10.1016/j.brat.2015.10.007. Epub 2015 Nov 2. PMID 26555157
- [Background] Moscovitch DA, Gavric DL, Merrifield C, Bielak T, Moscovitch M. Retrieval properties of negative vs. positive mental images and autobiographical memories in social anxiety: outcomes with a new measure. Behav Res Ther. 2011 Aug;49(8):505-17. doi: 10.1016/j.brat.2011.05.009. Epub 2011 May 26. PMID 21683343